CLINICAL TRIAL: NCT01475617
Title: Efficacy of a Novel Multivitamin-Mineral Supplement in Preventing Vitamin Deficiency in Postoperative Bariatric Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yasoo Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AQV-001
Record Dates: First submitted 2011-11-07; First posted 2011-11-21 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel Multivitamin/Mineral Supplement (Experimental): These subjects will be given a novel multivitamin/mineral supplement post RYGB bariatric surgery for 6 months duration.
  Interventions: Dietary Supplement: AquaVanta Chewable Tablet; Dietary Supplement: Nature Made Calcium Softgels
- Standard of care supplement (Active Comparator): These subjects will be given the standard recommended regimen at Johns Hopkins Bayview Medical Center post RYGB bariatric surgery for 6 months duration.
  Interventions: Dietary Supplement: Flinstones Complete; Dietary Supplement: Nature Made Calcium Softgels; Dietary Supplement: Twin Labs Iron Caps; Dietary Supplement: Rexall Vitamin B12 Tablet

INTERVENTIONS:
Dietary Supplement: AquaVanta Chewable Tablet — AquaVanta Chewable Tablet (proprietary formulation of vitamin and minerals) 2 times a day for 6 months
  Arms: Novel Multivitamin/Mineral Supplement
Dietary Supplement: Flinstones Complete — Flinstones Complete Multivitamin 2 times a day for 6 months
  Arms: Standard of care supplement
Dietary Supplement: Nature Made Calcium Softgels — Nature Made Calcium Softgels (Calcium Carbonate 600 mg and Vitamin D 200 mg) three times a day for 6 months
  Arms: Novel Multivitamin/Mineral Supplement
Dietary Supplement: Nature Made Calcium Softgels — Nature Made Calcium Softgels (Calcium Carbonate 600 mg and Vitamin D 200 mg) three times a day for 6 months
  Arms: Standard of care supplement
Dietary Supplement: Twin Labs Iron Caps — Twin Labs Iron Caps (Ferrous Fumarate) 18 mg per day for menstruating women for 6 months
  Arms: Standard of care supplement
Dietary Supplement: Rexall Vitamin B12 Tablet — Rexall Vitamin B12 Tablet (Cyanocobalamin 500 mcg)per day for 6 months
  Arms: Standard of care supplement

SUMMARY:
Approximately 33% of the US adult population can be classified as obese based on body mass index. This epidemic of obesity has resulted in over 200,000 bariatric surgeries performed every year for the treatment of "clinically severe obesity". Roux-en-Y gastric bypass (RYGB) is the most common bariatric procedure performed in the United States and has both restrictive and malabsorptive components. Despite the success of this procedure in creating long lasting weight loss, vitamin and iron deficiencies are common and can lead to significant morbidity if not appropriately addressed. Despite the American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery Medical Guidelines that include vitamin and mineral supplementation recommendations, there has been very little prospective research conducted to assess the efficacy and compliance of these micronutrient interventions.

This prospective randomized controlled clinical study will evaluate the efficacy of a novel vitamin/mineral supplement in decreasing micronutrient deficiencies in post operative bariatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 65 years of age
* Meet appropriate criteria for Roux-en-Y gastric bypass (RYGB) surgery as determined by the Principal Investigator at The John's Hopkins Center for Bariatric Surgery (JHCBS)

Exclusion Criteria:

* Allergy to a component of the formulations
* Recent (last 3 months) use of a dietary supplement other than a standard non-bariatric specific multivitamin supplement
* Documented levels of fat-soluble vitamins (A,D,E,K) or iron above the normal range
* Pregnant or lactating
* Expected poor compliance with medical regimen as assessed by JHCBS clinic care providers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plasma vitamin and mineral levels | 3 and 6 months compared to baseline

SECONDARY OUTCOMES:
Questionnaire regarding the palatability of the formulation and the ease of administration of the formats and dosing schedule | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Steele Steele, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The John's Hopkins Center for Bariatric Surgery (JHCBS), Baltimore, Maryland, United States

REFERENCES:
- [Derived] Perin J, Prokopowicz G, Furtado M, Papas K, Steele KE. A Randomized Trial of a Novel Chewable Multivitamin and Mineral Supplement Following Roux-en-Y Gastric Bypass. Obes Surg. 2018 Aug;28(8):2406-2420. doi: 10.1007/s11695-018-3177-0. PMID 29500675